CLINICAL TRIAL: NCT00888186
Title: Different Dyskinesias in Parkinson's Disease and Their Relation to Levodopa Pharmacokinetics
Acronym: DYSK-PD-2007
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish Parkinson's Disease Foundation (Unknown); Swedish Society for Medical Research (Other)
Responsible Party: Dag Nyholm, MD, PhD, Uppsala University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DYSK-PD-2007
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Parkinson Disease; Dyskinesias
Keywords: Dyskinesias; Duodenal levodopa infusion; Dose optimization; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1. Duodopa optimal dose (Active Comparator)
  Interventions: Drug: levodopa/carbidopa
- 2. Duodopa 20% too high dose (Experimental)
  Interventions: Drug: levodopa/carbidopa
- 3. Duodopa 10% too low dose (Experimental)
  Interventions: Drug: levodopa/carbidopa
- 4. Duodopa 20% too low dose (Experimental)
  Interventions: Drug: levodopa/carbidopa
- 5. Duodopa 10% too high dose (Experimental)
  Interventions: Drug: levodopa/carbidopa

INTERVENTIONS:
Drug: levodopa/carbidopa — intestinal gel, for continuous daytime infusion
  Other Names: Duodopa

SUMMARY:
The purpose of this study is to study different kinds of dyskinesias in advanced Parkinson's disease appearing at different levels of levodopa infusion dose. The hypothesis is that different dyskinesias (dystonia, chorea) correlate to different levels of levodopa concentrations, as detected in plasma.

DETAILED DESCRIPTION:
By using duodenal infusion of levodopa/carbidopa, the plasma concentration of levodopa can be kept fairly constant. Different doses, 10-20% higher or lower than the individually optimized dose will be used. Motor performance is captured by video recordings to be compared to/correlated with plasma levodopa concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Ongoing treatment with Duodopa
* Occurrence of dyskinesias, difficult to manage
* Age 30-90 years
* Hoehn & Yahr stage 3-5 at worst

Exclusion Criteria:

* Treatment with dopamine agonist or glutamate antagonist
* Dementia
* Psychosis
* Treatment with typical neuroleptics

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Correlation between plasma levodopa concentration and choreatic dyskinesia, dystonia, and parkinsonism | 3 days

SECONDARY OUTCOMES:
Correlation between choreatic dyskinesia, dystonia, and parkinsonism. | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Nyholm D, Nilsson Remahl AI, Dizdar N, Constantinescu R, Holmberg B, Jansson R, Aquilonius SM, Askmark H. Duodenal levodopa infusion monotherapy vs oral polypharmacy in advanced Parkinson disease. Neurology. 2005 Jan 25;64(2):216-23. doi: 10.1212/01.WNL.0000149637.70961.4C. PMID 15668416